CLINICAL TRIAL: NCT02109991
Title: A Prospective, Multi-center, Single-arm, Open-label Study Designed to Evaluate Safety, Tolerability and Performance Profile of the Colospan Device CG-100 in Patients Undergoing Colorectal Surgery
Brief Title: Safety, Tolerability and Performance Profile of the Colospan Device CG-100 in Patients Undergoing Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colospan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-001
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-07

CONDITIONS: Gastrointestinal Anastomosis

ARMS (1):
- CG-100 device (Experimental)
  Interventions: Device: CG-100 device

INTERVENTIONS:
Device: CG-100 device — Colorectal surgery performed per standard of care with deployment of the CG-100 device in the anastomosis site

SUMMARY:
The purpose of this study is to evaluate the CG-100 device, a single use, temporary intraluminal bypass device,intended to reduce contact of fecal content with an anastomotic site, following colorectal surgery (open or laparoscopic).

ELIGIBILITY:
Inclusion Criteria:

* The patient is scheduled to undergo an elective colorectal surgery (open or laparoscopic) which will require the creation of an anastomosis, maximally 20 cm proximal from the anal verge
* The patient is willing to comply with protocol-specified follow-up evaluations
* The patient signed Informed Consent

Exclusion Criteria:

* Pregnant or nursing female subjects
* Patient surgical treatment is acute (not elective)
* Patient has infections at the time of intervention
* Major surgical or interventional procedures within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study
* Patients with ASA (American Society of Anesthesiologists) classification > 3
* diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, local or systemic infection, ischemic bowel, carcinomatosis or extensively spread inflammatory bowel disease
* Patient is participating in another clinical trial within 30 days of screening
* Patient has been taking regular steroid medication in the last 6 months
* Contraindications to general anesthesia
* Patient has preexisting sphincter problems or evidence of extensive local disease in the pelvis
* Internal diameter lumen of the colon is smaller than 25 mm or larger than 34 mm
* Blood loss (> 500 cc)
* Leak test failure during surgery
* Any condition or surgical incidence where the device deployment can jeopardize the patient's safety or interferes with study outcome per the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events, and device related complications | During surgical procedure and up to 30 days (+/- 5)

SECONDARY OUTCOMES:
Occurrence of anastomotic leakage when the CG-100 is used | Up until device removal day (10 days +/-1)
Position of the device (internal sheath) | Device removal day (10 days +/-1)
Assessment of the device's application technique ease of placement and extraction of the device performance | Device removal day (10 days +/-1)
Determine subject tolerability of the device | Device removal day (10 days +/- 1)

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Gent, Ghent
- KBC Zagreb, Zagreb, Croatia
- Hungary (2):
  - Jahn Ferenc Hospital, Budapest
  - National Institute of Oncology, Budapest
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Rabin Medical Center, Petah Tikva
  - Assuta Medical Center, Tel Aviv